CLINICAL TRIAL: NCT03474692
Title: The Virta Health Registry for Remote Care of Chronic Conditions
Brief Title: Virta Health Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Virta Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-7
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Multiple Chronic Conditions; Chronic Disease; Disease Progression; Long-Term Care; Telemedicine
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this registry is to establish a research data repository, comprised of data generated in the course of providing clinical services to patients treated by Virta Health, to conduct secondary research on clinical interventions and chronic diseases.

DETAILED DESCRIPTION:
The purpose of this registry is to establish a research data repository, comprised of data generated in the course of providing clinical services to patients treated by Virta Health, to conduct secondary research on clinical interventions and chronic diseases.

The scope of research under this protocol includes the following:

1. Examining the effectiveness, safety, and sustainability of Virta Health clinical interventions for treating chronic diseases and prevention of or regression of associated adverse health outcomes.
2. Examining the cost-effectiveness and economic impact of Virta Health clinical interventions for treating chronic diseases and preventing or regressing associated adverse health outcomes.
3. Identifying demographics, clinical characteristics, comorbidities, concomitant treatments, genetic variants, and behavioral phenotypes that predict more or less favorable clinical outcomes of subjects to Virta Health clinical interventions for chronic diseases.
4. Examining the impact of mental health and the behavioral modification components of Virta Health clinical interventions on disease markers, comorbidities, and adverse health outcomes associated with Virta Health clinical interventions.
5. Characterizing typical presentation patterns, genetic determinants, biochemistry, and pathophysiology of the chronic diseases treated by Virta Health.
6. Exploring relationships between dietary composition and physiologic characteristics of chronic diseases.
7. Exploring the interrelationship and common clinical/biological features of the various chronic diseases under treatment by Virta Health.
8. Compiling case reports and case series of interesting disease presentations and outcomes, of the chronic diseases Virta Health treats, that may inform about the disease state and treatment responses.
9. Validating the integration of technological aids into Virta Health clinical interventions. Where the impacts of devices are examined, devices will be FDA-approved and approved, marketed devices. No safety data will be collected on devices; rather, research will focus only on the feasibility of adding the device to the treatment program, its relationship with participant behaviors and health outcomes, and patient satisfaction attributable to the device.
10. Understanding the relationships of patient needs, educational methods, and use of the Virta Health online Application, to subsequent patient satisfaction/clinical outcomes.

ELIGIBILITY:
Virta Health Patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving medical care from Virta Health for their chronic condition, most commonly type 2 diabetes, prediabetes, and metabolic syndrome.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2039-10 (Estimated); Study Completion 2039-10 (Estimated)

PRIMARY OUTCOMES:
Change in Chronic Disease Status | 6+ months
  change in disease status or markers of disease status over time

CONTACTS AND LOCATIONS:
Locations (1):
- Virta Health, Denver, Colorado, United States